CLINICAL TRIAL: NCT03953898
Title: The PRIME Trial: PARP Inhibition in IDH Mutant Effectiveness Trial. A Phase II Study of Olaparib in Isocitrate Dehydrogenase (IDH) Mutant Relapsed/Refractory Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: Using the Anticancer Drug Olaparib to Treat Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome With an Isocitrate Dehydrogenase (IDH) Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-03057; NCI-2019-03057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000027686; 10264 (Other: Yale University Cancer Center LAO); 10264 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia Post Cytotoxic Therapy; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity, or absence of remission after 6 cycles for patients without prior exposure to IDH inhibitors. Patients also undergo bone marrow aspiration and collection of blood throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Olaparib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial studies how well olaparib works in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory), or myelodysplastic syndrome. Patients must also have a change in the gene called the IDH gene (IDH mutation). Olaparib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of complete response (CR) to olaparib using a composite CR endpoint (CR + CR with incomplete hematologic response [CRi] + CR with partial hematologic response [CRh]) in subjects with isocitrate dehydrogenase (IDH)1/2 mutant myelodysplastic syndrome (MDS) or IDH1/2-mutant acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) to olaparib using a composite ORR endpoint (CR + morphologic leukemia-free state [MLFS] + partial response [PR]) in patients with IDH mutant AML or MDS treated with olaparib.

II. To establish the progression free survival (PFS) of patients with IDH mutant AML or MDS treated with olaparib.

III. To determine the overall survival (OS) of patients with IDH mutant AML or MDS treated with olaparib.

IV. To establish the duration of response (DOR) to treatment with olaparib. V. To evaluate the safety and tolerability of olaparib in AML or MDS patients.

EXPLORATORY OBJECTIVES:

I. To establish a relationship between treatment response and correlative studies such as plasma and bone marrow 2-hydroxyglutarate (2HG) levels, and IDH variant allele frequency.

II. To evaluate persistence of double strand breaks in IDH 1/2 mutant AML or MDS.

III. To evaluate response to therapy in the different IDH mutant genotypes.

IV. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES), ribonucleic acid (RNA) sequencing (RNAseq) order to:

IVa. Identify potential predictive and prognostic biomarkers beyond any genomic alteration by which treatment may be assigned.

IVb. Identify resistance mechanisms using genomic deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

V. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

VI. To bank blood and bone marrow aspirate obtained from patients at the EET Biobank at Nationwide Children's Hospital.

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity, or absence of remission after 6 cycles for patients without prior exposure to IDH inhibitors. Patients also undergo bone marrow aspiration and collection of blood throughout the study.

After completion of study treatment, patients are followed up at 90 days and then every 3 months until death.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of olaparib in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Diagnosis of MDS or AML per World Health Organization 2016 classification. AML may be de novo, or following a prior hematologic disorder, including MDS or Philadelphia chromosome-negative myeloproliferative neoplasm, and/or therapy-related.
* Patients must have a documented IDH1 or IDH2 mutation within 30 days of inclusion based on mutational testing. Only specific mutations that lead to a neomorphic phenotype will be eligible for enrollment, and include those listed below:

  * IDH1: R132V, R132G, R132S, R132L, R132C and R132H
  * IDH2: R140W, R140L, R140Q, R172W, R172G, R172S, R172M, R172K.
* Patients with AML or MDS should have disease that has relapsed after, or is refractory to, first-line therapy, with or without subsequent additional therapy.
* Patients with MDS should have at least a MDS-excess blasts (EB)1 at the inclusion and have a revised International Prognostic Symptom Score risk stratification of intermediate, high, or very high risk.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients may or may not have been previously treated with IDH targeted therapies.
* Patients who have undergone allogeneic stem cell transplant (alloSCT) are eligible if they are >= 180 days from stem cell infusion, have no evidence of graft versus host disease (GVHD) > grade 1, and are >= 2 weeks off all immunosuppressive therapy.
* Previous cytotoxic chemotherapy must have been completed at least 3 weeks and radiotherapy at least 2 weeks prior to Day 1 of treatment on the study, and all adverse events (AEs) (excluding alopecia) due to agents administered more than 4 weeks earlier should have recovered to < grade 1. Patients with hematologic malignancies are expected to have hematologic abnormalities at study entry. Hematologic abnormalities that are thought to be primarily related to leukemia are not considered to be toxicities (AEs) and do not need to resolve to < grade 1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky >= 60%).
* Patient must have recovered from toxicities of any prior treatment regimen (no Common Terminology Criteria for Adverse Events [CTCAE] grading over 1 for non-hematological toxicities, return to baseline for hematological values).
* Ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity may have a close relative, guardian, caregiver, or legally authorized representative consent on their behalf.
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) unless considered due to Gilbert's syndrome (measured within 28 days prior to administration of study treatment).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless considered due to organ leukemic involvement (measured within 28 days prior to administration of study treatment). If liver metastases are present in which case they must be =< 5 x ULN.
* Creatinine clearance of > 30 ml/min (measured within 28 days prior to administration of study treatment).
* Patients are eligible for this study if low blood count and transfusion support are due to the MDS/AML.
* Patients must have, in the best estimate of the treating physician, a life expectance of at least 12-16 weeks.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy).
* Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia.
* Patients with active central nervous system (CNS) leukemia or requiring maintenance intrathecal chemotherapy.
* Patients receiving concurrent chemotherapy, radiation therapy, or immunotherapy for AML/MDS.
* Patients actively receiving any other investigational agents.
* Management of treatment for patients with co-occurring mutations, like FLT3, will be prioritized by the treating physician after discussion of treatment options with the patient.
* Hyperleukocytosis with > 50,000 white blood cell (WBC)/mcl. Hydroxyurea for WBC count control is permitted before starting treatment and may be continued until day 28 of cycle 1. The maximum dose of hydrea will be 6 grams per day. Patients will be withdrawn from the study if > 50,000 WBC/mcl occur or recur > 14 days after starting treatment on the study.
* Active, uncontrolled infection. Patients with infection controlled with antibiotics are eligible.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients who are pregnant or nursing. Pregnant women are excluded from this study because olaparib is a PARP inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with olaparib, breastfeeding should be discontinued if the mother is treated with olaparib. These potential risks may also apply to other agents used in this study.
* Resting electrocardiogram indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT by Fridericia's formula (QTcF) prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Patients with symptomatic uncontrolled CNS disease. Imaging to confirm the absence of brain metastases is not required. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* The patient can receive a stable dose of corticosteroids, up to 20 mg by mouth (PO) prednisone daily, before and during the study as long as these were started at least 4 weeks prior to treatment.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Any previous treatment with PARP inhibitor, including olaparib.
* Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patient with active malignancies requiring active treatment that interferes with protocol therapy and/or with significant risk of clinical relapse within 12 months that would require treatment interfering with protocol therapy are excluded.
* Persistent toxicities (> Common Terminology Criteria for Adverse Event [CTCAE] grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment.
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks. Patients without reasonable alternative may be included in the trial after discussion with the medical monitor.
* Previous double umbilical cord blood transplantation (dUCBT).
* Breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2026-02-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rory M Shallis, Principal Investigator — Yale University Cancer Center LAO
Locations (11):
- United States (11):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Yale University, New Haven, Connecticut
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Olaparib): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity, or absence of remission after 6 cycles for patients without prior exposure to IDH inhibitors, or for up to 12 cycles. Patients also undergo bone marrow aspiration and collection of blood throughout the study.
  Biospecimen Collection: Undergo collection of blood
  Bone Marrow Aspiration: Undergo bone marrow aspiration
  Olaparib: Given PO
Period: Overall Study
Arm/Group | Treatment (Olaparib)
Started | 14
Started Therapy | 12
Completed | 0
Not Completed | 14
Not completed — Lack of Efficacy | 8
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 76 [42 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 10
  Race/Ethnicity: Latino | 2
  Race/Ethnicity: Asian | 1
  Race/Ethnicity: Black/African American | 0
  Race/Ethnicity: Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 14
ECOG PS [Count of Participants; unit: Participants] — ECOG Performance Status Scale (ECOG PS). ECOG PS ranks performance status on a scale of 0 to 5. 0 is "fully active" where 5 is "death".
  Participants
    0: Fully active | 3
    1: Unable to do strenuous activities | 9
    2: Able to walk and manage self-care | 2
    3: Confined to bed or a chair more than 50% of waking hours | 0
    4: Completely disabled | 0
    5: Death | 0
IDH mutation [Count of Participants; unit: Participants]
  IDH1 | 3
  IDH2 | 9
  IDH1 and IDH2 | 1
  MISSING | 1
Prior IDH inhibitor exposure [Count of Participants; unit: Participants]
  Yes | 8
  No | 6

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Overall Response Rate (ORR)
Description: Will be evaluated by Myelodysplastic Syndrome International Working Group (IWG) 2006 criteria (Cheson et al., 2006) and acute myeloid leukemia (AML) IWG 2003 criteria (Cheson et al., 2003) after 6 cycles of treatment. Cumulative ORR will include complete remission (CR), complete remission with incomplete blood count recovery (CRi), partial response (PR), and bone marrow complete remission (marrow CR) achieved at least at one point during these 6 cycles.
Time Frame: Up to 6 cycles
Population: Participants receiving treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 12
Participants
  Complete remission (CR) | 0
  Complete remission with incomplete hematologic response | 0
  Complete remission with partial hematologic response | 0
  Composite CR rate (CR+CRi+CRh) | 0
  No Response | 12

2. Secondary Outcome: ORR
Description: The effectiveness of the drug in patients for each cohort will be independently assessed by ORR. The exact two-sided 95% confidence intervals (CI) for the ORR will be reported. The CI based on the Greenwoods variance will be reported.
Time Frame: Up to 12 months
Population: Participants receiving treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 12
Participants
  OR = Yes | 0
  OR = No | 12

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on the Greenwoods variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease on the survival data. The adjusted p-values of the odds ratios and the adjusted 95% confidence interval will be reported.
Time Frame: From first day of therapy to the time of documentation of progression, death of any cause, or last follow-up, whichever comes first, assessed up to 12 months
Population: Participants receiving treatment
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 12
months | 2.3 [0.4 to 5.6]

4. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 3
Time Frame: From first day of therapy to the time of death or last follow-up, whichever comes first, assessed up to 12 months
Population: Participants receiving treatment
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 12
months | 3.4 [0.4 to 35.3]

5. Secondary Outcome: Duration of Response (DOR)
Time Frame: From first documentation of response to the time of documentation of progression, death of any cause, or last follow-up, whichever comes first, assessed up to 12 months
Population: no patients responded to treatment
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Adverse Events
Description: Non-hematologic toxicity will be evaluated by Common Terminology Criteria for Adverse Events version 5 criteria. Presented are the count of those that experienced at least one non-serious adverse event.
Time Frame: Up to 12 months
Population: 12 pariticipants received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 12
Participants | 12

7. Other Pre Specified Outcome: Change in 2-hydroxyglutarate (2HG) Levels
Description: The Mann-Whitney U test will be used to test for differences in post-treatment plasma 2HG concentrations between patients with a response to treatment and those without. Will also test for differences in Delta2HG (defined as pre-treatment minus post-treatment plasma concentration) between patients with a response to treatment and those without. Differences with p =< 0.05 will be considered significant. The area under the receiver operating characteristic curve (ROC AUC) will be calculated to determine the cutoff value of the Delta2HG difference. The optimal cutoff value will be determined at the point on the ROC curve at (sensitivity + specificity - 1) is maximized.
Time Frame: Up to 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Assessment
Description: Will define MRD based on the variation of the variant allele frequency of the IDH1/2 mutation in the bone marrow of the patients before and during therapy. Will evaluate two different variables: MRD negativity (defined by the absence of detection of the IDH mutant in the sample) and the molecular response (defined by the log reduction of the frequency of the mutant allele). MRD negativity is a qualitative variable and will be reported as a percentage with 95% confidence interval for each time point and mutation. Will compare the different groups using a Chi-Square test. Molecular response is a quantitative variable reported as a median, min and max for each time point and we will use a student t test for the comparison of the different groups.
Time Frame: Up to 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mutant Allele Frequency
Description: Will be estimated using Poisson distribution model as the fraction of positive reads divided by total reads containing a target. The limit of detection will be defined for each mutation as the mean value of IDH1/2 wild-type controls plus three standard deviations.
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Median time from 1st dose to off-study: 74.5 days
Arm/Group | Treatment (Olaparib)
All-Cause Mortality (participants affected / at risk) | 10/12
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Olaparib) (N=12)
Constipation (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Dyspnea (Investigations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Fungemia (Infections and infestations) | 1
Hypoxia (Investigations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 4
Mucositis oral (Gastrointestinal disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Respiratory failure (Investigations) | 2
Sepsis (Infections and infestations) | 4
Sinus tachycardia (Cardiac disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Olaparib) (N=12)
Anemia (Blood and lymphatic system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Vision decreased (Eye disorders) | 1
Disease progression (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Neck edema (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Infections & infestations - Other - Sepsis (Infections and infestations) | 3
Lung infection (Infections and infestations) | 3
Skin infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Cytomegalovirus infection reactivation (Infections and infestations) | 1
Fungemia (Infections and infestations) | 1
Infections & infestations - Other - Covid-19 (Infections and infestations) | 2
Lip infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 3
White blood cell decreased (Investigations) | 3
ALT increased (Investigations) | 2
AST increased (Investigations) | 2
Activated PTT prolonged (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Investigations - Other, specify - Night Sweat (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms - Other - Adrenal Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms - Other - Lung Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Skin & subcutaneous tissue -Other - Cellulitis (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT03953898/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT03953898/ICF_001.pdf